CLINICAL TRIAL: NCT05992324
Title: A Validation Study to Evaluate the Performance of Caption Health Lung Guidance and Interpretation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caption Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LungPivotal
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Shortness of Breath
Keywords: Lung Ultrasound; B-Lines; POCUS by non-expert user
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patients presenting with clinical suspicion of B-Lines (Experimental): Patients will undergo two 8-zone protocol lung ultrasound exams. One exam will be conducted by an expert lung ultrasound user without Caption LungAI and will last approximately 5-10 minutes. The second exam will be conducted by a healthcare professional with Caption LungAI and will last approximately 15-20 minutes.
  Interventions: Device: Caption LungAI

INTERVENTIONS:
Device: Caption LungAI — Caption LungAI is a software that is designed to help non-expert healthcare professionals acquire diagnostic quality images on an 8-zone lung protocol for both healthy patients and patients presenting with pathology such as B-Lines.

SUMMARY:
The purpose of this study is to assess the efficacy of Caption LungAI.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo two 8-zone protocol lung ultrasound exams. One exam will be conducted by an expert lung ultrasound user without Caption LungAI and one exam conducted by a (non-expert) healthcare provider who is trained on Caption LungAI and will use Caption LungAI to capture images.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients presenting to the hospital or outpatient setting with shortness of breath and suspected B-lines.

Exclusion Criteria:

* Patients in extremis/in whom a research lung ultrasound would not normally be performed due to other priorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Image Quality (Trained Healthcare Professional) | Up to 24 weeks from completion of the study.
  Evaluate the product's ability to assist the user to capture a LUS image with diagnostic quality. Percentage of zones with diagnostic image quality > 0.80
B-Lines Detection | Up to 24 weeks from completion of the study.
  Evaluate the product's ability to retrospectively detect present B-lines on images acquired by a local expert with no Caption Lung AI assistance. AUROC > 0.80; Sensitivity (Se) > 0.80; Specificity (Sp) > 0.75
B-Line Significance | Up to 24 weeks from completion of the study.
  Evaluate the product's ability to retrospectively detect B-lines of significant severity on images acquired by a local expert with no Caption Lung AI assistance. AUROC > 0.80; Sensitivity (Se) > 0.80; Specificity (Sp) > 0.75
Remote Reader Performance | Up to 24 weeks from completion of the study.
  Evaluate the product's impact on a remote expert reader's ability to interpret LUS images. Difference Between Aided &
  Unaided Groups:
  AUROC > 0.00; Sensitivity (Se) > 0.00; Specificity (Sp) > 0.00

SECONDARY OUTCOMES:
Sub-group Analyses | Up to 24 weeks from completion of the study.
  The following sub-group analyses will be performed for the primary endpoints: age (< 65, ≥ 65), BMI group (< 25, 25 ≤ BMI < 30, ≥ 30), gender (Male / Female), site location, trained HCP, and zone of the image (1 - 8).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The Moses H. Cone Memorial Hospital, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baloescu C, Bailitz J, Cheema B, Agarwala R, Jankowski M, Eke O, Liu R, Nomura J, Stolz L, Gargani L, Alkan E, Wellman T, Parajuli N, Marra A, Thomas Y, Patel D, Schraft E, O'Brien J, Moore CL, Gottlieb M. Artificial Intelligence-Guided Lung Ultrasound by Nonexperts. JAMA Cardiol. 2025 Mar 1;10(3):245-253. doi: 10.1001/jamacardio.2024.4991. PMID 39813064